CLINICAL TRIAL: NCT01750645
Title: Management of the Idiopathic Overactive Bladder With Intradetrusor Injection of Type-A Botulinum Toxin: Systematic Review of the Literature
Brief Title: Management of the Idiopathic Overactive Bladder With Botulinum Toxin: Systematic Review
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clínica Infantil Colsubsidio (Other)
Responsible Party: Principal Investigator, Hugo Enrique López, MD, MD, Clínica Infantil Colsubsidio
Other Study IDs: COLS-201207
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention Group
  Interventions: Drug: Intradetrusor Injection of Type-A Botulinum Toxin
- Control Group
  Interventions: Other: Other interventions analyzed according to protocol

INTERVENTIONS:
Drug: Intradetrusor Injection of Type-A Botulinum Toxin
  Groups: Intervention Group
Other: Other interventions analyzed according to protocol — * Placebo
  * Different dosage of Type-A Botulinum Toxin injected
  * Anticholinergic drugs
  Groups: Control Group

SUMMARY:
Overactive bladder is defined as a syndrome composed of urgency, increased urinary frequency, and sometimes urinary incontinence; its etiology may be characterized as neurogenic or non-neurogenic (i.e., idiopathic). This illness has a great impact in quality of life and one of the available treatments is the injection of Botulinum Toxin. This study aims to review the efficacy and safety of type-A Botulinum Toxin in the management of Idiopathic Overactive Bladder. A systematic search was performed in MEDLINE, EMBASE, CENTRAL and LILACS, and the controlled randomized clinical trials were chosen to review with the CONSORT criteria by independent reviewers. Outcomes analyzed were the efficacy of the intervention for relieving the symptoms (urgency, frequency and urgency incontinence), adverse events to treatment, change in quality of life and urodynamic measures.

ELIGIBILITY:
Inclusion Criteria:

* Controlled randomized clinical trials
* Adult patients diagnosed with idiopathic overactive bladder
* Language of the study: english

Exclusion Criteria:

* Diagnosis of neurogenic overactive bladder
* Patients under 18 years old
* Use of Type-B Botulinum Toxin as the intervention
* Other types of studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with idiopathic overactive bladder
Sampling Method: Non-Probability Sample
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the intervention for relieving the symptoms (urgency, frequency and urgency incontinence) | Minimun follow-up period of 12 weeks

SECONDARY OUTCOMES:
Adverse events to treatment (urinary retention and urinary tract infections) | Minimun follow-up period of 12 weeks
Change in quality of life | Minimun follow-up period of 12 weeks
Change in urodynamic measures | Minimun follow-up period of 12 weeks
  Increase in maximum cystometric capacity, first desire to void, normal desire to void, postvoid residual volume, and the presence/abscence of detrusor overactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo E López, MD, Principal Investigator — Clínica Infantil Colsubsidio
Locations (1):
- Clínica Infantil Colsubsidio, Bogotá DC, Bogotá DC, Colombia